CLINICAL TRIAL: NCT02142101
Title: Gut Microbiota of Renal Patients
Brief Title: Evaluation of Gut Bacteria in Patients With Polycystic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 13-1798
Record Dates: First submitted 2014-05-07; First posted 2014-05-20 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Polycystic Kidney Disease
Keywords: Gut Microbiota; Polycystic kidney disease; Chronic kidney disease; Uremic metabolites
MeSH Terms: conditions — Polycystic Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum and urine will be saved for metabolite analysis; stool will be used to extract bacterial DNA for sequencing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- GFR >60: 5 patients with polycystic kidney disease with eGFR > 60 ml/min.
- GFR 15-60: 5 patients with polycystic kidney disease with eGFR between 15-60 ml/min.
- GFR <15: 5 patients with polycystic kidney disease with eGFR <15 ml/min.

SUMMARY:
Gut microbes can influence numerous aspects of human biology. Alterations in the function and composition of gut microbial flora (gut microbiota ) have been linked to inflammatory bowel disease, chronic inflammation, dyslipidemia, diabetes mellitus, atopic disorders, cardiovascular disease, neoplasms, and obesity. However, little is known whether renal failure alters the composition of gut microbiota and whether an alteration in the gut microbiota of patients with renal failure impacts on the development of co-morbid conditions such as accelerated atherosclerosis, abnormal bone mineral metabolism, and chronic inflammation that are associated with renal failure. Nonetheless, several lines of evidence suggest that renal failure alters the chemical environment of the intestinal lumen, which could impose a selective pressure on the growth of certain gut microbes. The investigators hypothesize that the gut microbiota of patients with renal failure is different from those without renal failure. To test this hypothesis the investigators are conducting a cross-sectional study of gut microbiota in patients with different degrees of renal failure due to polycystic kidney disease (PKD).

DETAILED DESCRIPTION:
Studies have shown that gut microbes can influence numerous aspects of human biology, and alterations in the function and composition of gut microbial flora (microbiota) play a major role in the pathogenesis of diverse human illnesses such as chronic inflammation, diabetes mellitus, and cardiovascular diseases. Gut microbes provide protection against pathogenic organisms, contribute to energy metabolism, serve a clear role in the development and modulation of the human gut immune system, and participate in nitrogen and micronutrient homeostasis by synthesizing amino acids and various vitamins. However, whether the composition of gut microbes is altered in human with renal failure has not been clearly demonstrated. Furthermore, whether alterations in the gut microbiota due to renal failure contribute to development of co-morbid conditions associated with CKD has never been examined. There are several lines of evidence to suggest that the gut microbiota is likely altered in patients with CKD. It has been established that protein assimilation in the small intestine is impaired in CKD .

To examine the impact of renal failure on the composition of gut microbiota we are studying patients with renal failure due to polycystic kidney disease (PKD). PKD is the fourth leading cause of kidney failure, and is the most common genetic kidney disease. Compared to patients with renal failure due to diabetic nephropathy, hypertension, and glomerulonephritis, patients with PKD have virtually no major co-morbid medical conditions or associated medical interventions (i.e. antimicrobial or anti-inflammatory therapies) that could potentially alter the gut microbiota, and confound the interpretation of data.

Objectives

1. To compare the gut microbiota in fecal samples of PKD patients with different degrees of renal disease.
2. To determine whether alteration in the composition of gut microbiota is linked to serum levels of metabolites and uremic solutes that are known to be associated with symptoms of uremia.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Patients with PKD.
* Patients are able to understand and give consent.

Exclusion Criteria:

* Patient on antibiotics or vitamin supplement (except vitamin D analogs) in the last three months.
* Advanced liver disease, advanced cardiovascular disease, heart failure with EF < 30%, and autoimmune disease.
* The use of chemotherapy, antibiotics, immunosuppressive medications, probiotics, and steroid in the last three month.
* Intravenous or oral iron supplementation, laxatives, and kayexalate in the last month.
* History of intra abdominal surgery, small or large intestine resection or small bowel obstruction.
* History of colon cancer or gastrointestinal bleed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: o All subjects with diagnosis for cystic kidney disease, who were evaluated at Mount Sinai Hospital, Renal clinic, Internal Medicine Associates clinic and Faculty Practice Associates clinics will be identified via the electronic medical system (EPIC).
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Microbiome sequencing and diversity and its correlation with renal function | at 2 weeks
  The diversity of gut bacterial population and its correlation with the renal function, bacterial DNA extract will be sequenced using MiSeq. Data will be analyzed using QiiMe program.

SECONDARY OUTCOMES:
Uremic metabolites and its correlation with gut microbiota | at 2 weeks
  To evaluate the uremic metabolites and its association with specific bacterial phylum identified by bacterial DNA sequencing
Kidney function and uremic metabolites | at 2 weeks
  To evaluate the correlation of uremic metabolites in urine and its correlation with renal function by analyzing non-targeted metabolite profiling platform.
Vit D level | at 2 weeks
  The correlation of Vit D level with gut bacterial population, and its effects on urine and serum metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: John C He, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States